CLINICAL TRIAL: NCT02120703
Title: Gabapentin vs. Pregabalin for Post Operative Pain in Lumbar Microdiscectomy: a Randomized Controlled Trial.
Brief Title: Pregabalin Compared to Gabapentin for Pain Control in Lumbar Disc Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ghulam Murtaza, Dr., Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 173-SUR-ERC-10
Record Dates: First submitted 2014-04-19; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Intervertebral Disc Prolapse
Keywords: Pregabalin; gabapentin; microdiscectomy; pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain | interventions — Pregabalin; Gabapentin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gabapentin (Active Comparator)
  Interventions: Drug: Gabapentin
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregablin 75 mg per oral two times a day
  Arms: Pregabalin
Drug: Gabapentin — Gabapentin 200 mg twice daily per oral
  Arms: gabapentin

SUMMARY:
Pregabalin is claimed to have superior analgesic effect at lower doses and better pharmacological profile as compared to gabapentin esp. in perioperative pain control after major surgeries like intervertebral disc surgery.

The investigators found that pregabalin is equivalent to gabapentin for relief of post-operative pain at a lower dose in patients undergoing intervertebral disc surgery.

ELIGIBILITY:
Inclusion Criteria:

* 30-60 years age
* Any gender
* elective micro discectomy for intervertebral disc prolapse

Exclusion Criteria:

1. micro discectomy at two or more vertebral levels,
2. Instrumentation i.e. pedicle screw fixation, hooks etc.,
3. history of steroids or alcohol use,
4. Multiple co-morbids i.e. renal failure, chronic liver disease,
5. use of anticonvulsant drugs,
6. Spinal deformity,
7. Obesity (BMI >30), 8) inability to understand and respond VAS and

9) patients with known allergy to GABA analogues.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain | 7 days
  Pain measurement using Visual Analogue Score at 24 hours and 7th day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Qadeer, FCPS, Principal Investigator — The Aga Khan University Hospital, Karachi, Pakistan
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan